CLINICAL TRIAL: NCT05947019
Title: Efficacy and Safety of Low-Level Monochromatic Red-Light for High Myopia Control in Adults: A Randomized, Controlled, Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Low-Level Monochromatic Red-Light for High Myopia Control in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QX-2022-A-014
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: High Myopia
Keywords: High Myopia; LLLT; Adults
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Red-Light threapy plus glasses threapy (Experimental): Myopic amblyopia comprehensive treatment equipment + conventional optometry with glasses for treatment
  Interventions: Device: Myopic amblyopia comprehensive treatment instrument; Device: Glasses
- glasses threapy (Experimental): conventional optometry with glasses for treatment
  Interventions: Device: Glasses

INTERVENTIONS:
Device: Myopic amblyopia comprehensive treatment instrument — Myopic amblyopia comprehensive treatment instrument is produced by Suzhou Industrial Park Zuoguan Medical Equipment Co., LTD.
  Arms: Low-Level Red-Light threapy plus glasses threapy
Device: Glasses — Optometry with glasses as a routine treatment

SUMMARY:
The purpose of this clinical study is to confirm the effectiveness and safety of low-level monochromatic red-light for high myopia control in adults

DETAILED DESCRIPTION:
Currently, there is still a lack of effective methods for managing adult high myopia globally. The Elsing Myopia and Amblyopia Therapy Instrument, developed by Suzhou Industrial Park Zuoguan Medical Equipment Co., Ltd., has gained widespread usage in mainland China for amblyopia treatment and myopia control. This instrument utilizes low-intensity laser therapy (LLLT) for treatment, demonstrating improvements in visual acuity without any local or systemic side effects. The low-intensity laser induces photochemical reactions in the retina, such as enhancing cytochrome C oxidase activity, modulating gene expression to regulate the mitochondrial respiratory chain, and increasing the biological activity of nitric oxide. These mechanisms have been applied in the treatment of age-related macular degeneration and diabetic retinopathy. As the onset of myopia is closely linked to retinal signaling pathways, preliminary test data suggests that the instrument can significantly slow down myopia progression. This study aims to investigate the potential of low-intensity laser therapy in preventing and treating high myopia in adults, providing innovative approaches to mitigate the widespread impact of high myopia.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 40 years, regardless of gender.
2. Presence of myopic refractive error in at least one eye, with myopic lens power after mydriasis exceeding 6.00D, diffusivity less than 2.00D, binocular anisometropia less than 3.00D, and best corrected distance visual acuity of at least 0.6, as well as near visual acuity of at least 0.6.
3. Normal cognitive abilities and language communication skills, capable of actively cooperating with the required treatment.
4. Absence of contraindications for atropine use, such as acute ocular inflammation, dry eye, keratoconus, and diabetes.
5. Written informed consent obtained from the patients.

Exclusion Criteria:

1. History of photoallergy, glaucoma, trichiasis syndrome, ocular hypertension, fundus macula lesions, or eye injuries.
2. Corneal curvature examination revealing an average K value of the anterior corneal surface of ≥45.
3. Presence of systemic diseases (e.g., heart, liver, kidney diseases) and congenital hereditary myopia.
4. Chronic eye diseases, including ocular trauma, strabismus, or previous ocular surgery, as well as allergic conjunctivitis.
5. Previous internal trichiasis, severe corneal opacity, conjunctival infection, or other eye diseases.
6. Neurological diseases, allergies, or contraindications to atropine or other therapeutic drugs.
7. Presence of immune system and systemic diseases such as albinism, psoriasis, nephrotic syndrome, systemic lupus erythematosus, or diabetes.
8. Epilepsy or mental disorders that hinder normal communication.
9. Previous use of other treatments to control myopia progression, such as anticholinergic drugs like atropine within the past 3 months, or participation in other studies involving functional frame lenses, multifocal soft lenses, or similar interventions.
10. Any other situation deemed unsuitable for participation in the study by the researcher.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in axial length of the left and right eyes | baseline, 30days, 90 days, 180 days
  The axis of the eye was assessed utilizing the IOL Master (version 5.02, Carl Zeiss, Jena, Germany), which employed simulated eye calibration prior to measurements. To ensure accuracy, three consecutive measurements were taken, and the average value was obtained. If the difference between any two measurements exceeded 0.05mm, a re-measurement was performed.

SECONDARY OUTCOMES:
Changes of equivalent spherical mirror after mydriatic optometry | baseline, 180 days
  Based on previous experience, this instrument requires a treatment duration of 180 days to demonstrate its preventive and control effects. Therefore, the 180-day data changes will be utilized as the evaluation indicator.

CONTACTS AND LOCATIONS:
Overall Officials: He Jiangnan, PhD, Study Director — Shanghai Eye Disease Prevention & Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No